CLINICAL TRIAL: NCT01336452
Title: Noninvasive Surrogate Marker for Advanced Hepatocellular Carcinoma Response to Concurrent Chemoradiotherapy: MR Perfusion, Contrast Enhanced Ultrasound and Biomarkers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2010-0566
Record Dates: First submitted 2011-04-13; First posted 2011-04-15 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Advanced Adult Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CCRTx (Other): consecutive patients who plan to undertake CCRTx due to advanced hepatocellular carcinoma
  Interventions: Radiation: DCE MRI

INTERVENTIONS:
Radiation: DCE MRI — DCE (dynamic contrast enhanced) MRI will be obtained just before CCRTx and immediately after finishing CCRTx with 0.1mmol/kg of MR contrast media; CEUS will be obtained just before CCRTx, immediately after finishing CCRTx, and 1 month after CCRTx with 2.4 mL of SonoVue. Blood sampling for biomarker analysis will be performed just before CCRTx, immediately after finishing CCRTx, and 1 month after CCRTx (20mL)

SUMMARY:
Hepatocellular carcinoma is the sixth most common malignancy and the third most common cause of cancer-related death worldwide. The incidence of HCC is rising in Europe and the United States and is expected to continue to increase during the next 2 to 3 decades. The expected survival rate is still decimal, especially in patients with advanced HCC. However, in recent years, several treatment methods for patients with advanced HCC, including antiangiogenic chemotherapy, radiotherapy, concurrent chemoradiotherapy, and DC bead transarterial chemoembolization, have been developed. Among these new treatment methods, concurrent chemoradiotherapy has also proved to increase patient's survival rate. It is important to predict treatment response before treatment or immediately after treatment because there are several other treatment options as mentioned above. Recently, there have been several reports that MR perfusion parameters such as Ktrans can predict treatment response in cervical cancer and colorectal cancer. Therefore the purpose of the investigators study is to evaluate the feasibility of predicting treatment response by MR perfusion, contrast enhanced ultrasound parameters and biomarkers (IL-6, IL-12 and VEGF) in patients with advanced hepatocellular carcinoma who undertake concurrent chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have advanced hepatocellular carcinoma and plan to undertake concurrent chemoradiotherapy.
* Patients willing to undergo the study procedure
* Patients who are fully informed about the study and have signed the informed consent form

Exclusion Criteria:

* Patients (men or women) under 20 years of age
* Patients who have been received any other treatment including TACE, operation, TACI, systemic chemotherapy, intraarterial chemotherapy, antiangiogenic therapy
* Patients who have hypersensitivity to MR or US contrast agents
* Women who are pregnant, lactating or who are of childbearing potential and have not had a negative pregnancy test at baseline visit
* Patients not eligible to contrast media injection according to product labeling
* Patients with a contraindication for MRI or CT
* Patients with impaired renal function (e.g. acute renal failure) or patients on dialysis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
characteristic of Perfusion MR | 1 month
  Ktrans (volume transfer constant between the EES and the blood plasma), Kep (rate constant between the EES and the blood plasma), Ve (Ktrnas/Kep: EES fractional volume), tumor volume

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea